CLINICAL TRIAL: NCT05045222
Title: ECOST = Economic and Clinical Outcomes of (Whole Exome) Sequencing in Tapestry
Brief Title: Economic and Clinical Outcomes of (Whole Exome) Sequencing in Tapestry
Acronym: ECOST
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-010400
Record Dates: First submitted 2021-07-28; First posted 2021-09-16 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Health Care Utilization
Keywords: Tapestry; Quality of life - adjusted life years; ECOST
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to learn more about the impact of genetic testing on healthcare costs, clinical care, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Tapestry patients who have received genetic results, regardless of positive or negative testing results.
* Age of 18 and older.
* Patients with an established Mayo Clinic provider prior to their enrollment in Tapestry.

Exclusion Criteria:

* Individuals less than 18 years old.
* Patients without capacity to consent (i.e., needing legal authorized representatives).
* Prisoners.
* Subjects eligible for chart review, without a Minnesota Research Authorization on record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include participants of the Tapestry study, which is an ongoing project aimed at studying the genetic risk factors that impact medical care of patients at Mayo Clinic. This study will include the first 15,000 Tapestry patients who received results of 11 genes (incidental findings) after undergoing WES using a saliva sample and were enrolled January 2020 onwards. Chart review of up to 85,000 records will accompany the 15,000 enrolled and completing surveys for a total of 100,000 accrued.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2031-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life measured through adjusted years. | Every 12 months for 5 years after enrollment.
  Measuring quality of life through adjusted years due to learning Tapestry test results.
Disease incidence measured by disease count per 100 participants. | 12 months
  Number of disease incidences per 100 participants.
Change in utilization measured by total number of office visits, hospital stays, ER visits, and length of visits. | Every 12 months for 5 years after enrollment.
  Composite of: Number of Office-based visits. Number of Hospital stays and length of visits. Number of ER visits.
Change in costs measured by disease related and all-cost related costs. | Every 12 months for 5 years after enrollment.
  Cost Composite of: Disease-related costs. Disease-related costs by utilization category. All-cause costs. All-cause costs by utilization category.

SECONDARY OUTCOMES:
Change in quality of life measured through adjusted years from subgroups. | Every 12 months for 5 years after enrollment.
  Measuring quality of life through adjusted years due to learning Tapestry test results categorized by subgroups: minority races, 65 years and older, etc.
Change in quality of life measured through adjusted years from different scenarios. | Every 12 months for 5 years after enrollment.
  Measuring quality of life through adjusted years due to learning Tapestry test results categorized by different scenarios: disease comorbidities, patient income, education, adherence to medical orders, etc.
Disease incidence from subgroups. | 12 months
  Number of disease incidences per 100 hundred participants categorized by subgroups: minority races, 65 years and older, etc.
Disease incidence from different scenarios.. | 12 months
  Number of disease incidences per 100 hundred participants categorized by different scenarios: disease comorbidities, patient income, education, adherence to medical orders, etc.
Change in utilization from subgroups. | Every 12 months for 5 years after enrollment.
  Composite of: Number of Office-based visits. Number of Hospital stays and length of visits. Number of ER visits. All categorized by subgroups: minority races, 65 years and older, etc.
Change in utilization from different scenarios. | Every 12 months for 5 years after enrollment.
  Composite of: Number of Office-based visits. Number of Hospital stays and length of visits. Number of ER visits. All categorized by different scenarios: disease comorbidities, patient income, education, adherence to medical orders, etc.
Change in costs from subgroups. | Every 12 months for 5 years after enrollment.
  All-cause costs. All-cause costs by utilization category. All categorized by subgroups: minority races, 65 years and older, etc.
Change in costs from different scenarios. | Every 12 months for 5 years after enrollment.
  All-cause costs. All-cause costs by utilization category. All categorized by different scenarios: disease comorbidities, patient income, education, adherence to medical orders, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Niloy Jewel Samadder, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials